CLINICAL TRIAL: NCT00786539
Title: Investigation of the Nature and Prevalence of Mitochondria Disease
Brief Title: Mitochondria Inborn Errors of Metabolism and ANT Defects in Mitochondria Diseases
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Virginia Kimonis, MD, MRCP, University of California, Irvine
Other Study IDs: 20022608
Record Dates: First submitted 2008-11-04; First posted 2008-11-06 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Mitochondrial Disease
Keywords: mitochondrial
MeSH Terms: conditions — Mitochondrial Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Diffuse Optical Spectroscopy — mitochondria

SUMMARY:
The objective of this research protocol is to continue investigation of the nature and prevalence of mitochondria disease and to aid patients and health care providers in the understanding of these complex disorders.

This research study brings together many clinical sub-specialists to address the etiology of these disorders and to develop more effective approaches for their diagnoses and more reliable prognoses.

DETAILED DESCRIPTION:
The non-invasive device named Diffuse Optical Spectroscopy developed at the Beckman Laser Institute is to be used to measure various physiological parameters. Since mitochondria produce most of the energy necessary for cellular function, their efficacy is most important for systems with a high energy demand like the brain, heart, skeletal muscle, kidney, liver, and endocrine tissues. As a result, mitochondria diseases usually manifest as complex, multi-organ disorders, requiring multispecialty investigations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female all ages group with diagnosis of mitochondrial disorder

Exclusion Criteria:

* Subjects with visual, auditory and/or neurological problems known to result from toxic or environmental effects

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population with mitochondrial disorder and/or their relatives will be referred to MITOMED by Primary Care Physicians or by Clinical Specialists.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2006-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Symptoms of Mitochondrial diseases | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bruce J Tromberg, PhD, Principal Investigator — Beckman Laser Institute University of California Irvine; Virginia Kimonis, MD, Principal Investigator — UCIMC Pediatrics
Locations (1):
- Beckman Laser Institute Medical clinic, Irvine, California, United States